CLINICAL TRIAL: NCT02357628
Title: Effect of Regulated Oxygen-Enriched Negative Pressure Therapy (RO-NPT) On Soft Tissue Wound Repair
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0078-14-HYMC
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Wounds and Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Research Group I: Wound treatment with RO-NPT 40%
  Interventions: Device: Wound treatment with RO-NPT
- Research Group II: Wound treatment with RO-NPT 60%
  Interventions: Device: Wound treatment with RO-NPT
- Research Group III: Wound treatment with RO-NPT 40% and irrigation
  Interventions: Device: Wound treatment with RO-NPT; Device: Wound Irrigation

INTERVENTIONS:
Device: Wound treatment with RO-NPT
  Other Names: Oxygen-enriched vacuum therapy
Device: Wound Irrigation
  Groups: Research Group III

SUMMARY:
The investigators believe that regulated oxygen-enriched negative Pressure Therapy (RO-NPT) will be beneficial in the reduction or elimination of anaerobic infection in hard-to-heal soft tissue wounds.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hard-to-heal wounds

Exclusion Criteria:

* Everyone else

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients presenting at the Hillel Yaffe Medical Center for treatment of hard-to-heal wounds that have been selected for RO-NPT.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Wound Closure | One Month
  Before treatment and after treatment wound area measurements will indicate percentage of closure

CONTACTS AND LOCATIONS:
Overall Officials: Moris Topaz, MD, Phd, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel